CLINICAL TRIAL: NCT03539640
Title: The Effects of Positive End-expiratory Pressure on the Position, Length and Contractibility of the Diaphragm.
Brief Title: Effect PEEP on Diaphragm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof.dr. L.M.A. Heunks, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NL63905.029.17
Record Dates: First submitted 2018-04-17; First posted 2018-05-29 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Diaphragm Disease
Keywords: PEEP; Diaphragm

STUDY DESIGN:
Intervention Model Description: All participants will receive the same protocol with different levels of PEEP ventilation during the first part of the study (physiological part), so the interventional study model for this part is single group. During the second part (MRI), participants are randomized for one of the three available PEEP levels (5, 10 or 15 cmH2O), so the study model for this part is parallel.
Who Masked: Outcomes Assessor
Masking Description: The assessor of the MRI measurements will analyze the MRI data in a blinded fashion. The rest of the outcomes will not be analyzed in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEEP level of 5 cmH2O (Active Comparator): During second part of the study (MRI) Diaphragm position
  Interventions: Other: PEEP: 5 cmH2O
- PEEP level of 10 cmH2O (Active Comparator): During second part of the study (MRI) Diaphragm position
  Interventions: Other: PEEP: 10 cmH2O
- PEEP level of 15 cmH2O (Active Comparator): During second part of the study (MRI) Diaphragm position
  Interventions: Other: PEEP: 15 cmH2O

INTERVENTIONS:
Other: PEEP: 5 cmH2O — During second part of the study (MRI)
  Arms: PEEP level of 5 cmH2O
Other: PEEP: 10 cmH2O — During second part of the study (MRI)
  Arms: PEEP level of 10 cmH2O
Other: PEEP: 15 cmH2O — During second part of the study (MRI)
  Arms: PEEP level of 15 cmH2O

SUMMARY:
This study evaluates the effect of positive end-expiratory pressure on the position, length and function of the diaphragm. During the first part of the study, physiological measurements of the diaphragm will be performed while participants receive non-invasive ventilation at different PEEP levels. During the second part of the study, MRI measurements of the diaphragm will be performed during a change in PEEP level.

DETAILED DESCRIPTION:
In almost all mechanically ventilated patients, positive end-expiratory pressure (PEEP) is used. Its function is to prevent alveolar collapse and to maintain oxygenation. However, it has recently been found that PEEP may contribute to diaphragm weakness, which is an important problem in the intensive care unit (ICU). This study showed that mechanical ventilation with PEEP resulted in a caudal displacement of the diaphragm, since PEEP increases the end-expiratory volume. Furthermore, their study in rats showed that this displacement resulted in a reduced fiber length and sarcomere length on the short term.

After rats were ventilated with PEEP for 18 hours, it was found that adaptation of the diaphragm occurred; i.e. the number of sarcomeres were decreased. It is hypothesized that this adaptation may also occur in mechanically ventilated patients. This could lead to problems in weaning a patient off the ventilator, as PEEP is abruptly removed during a spontaneous breathing trial (SBT). This leads to a reduction in end-expiratory volume which would mean that the newly-adapted diaphragm fibers are being stretched. These stretched muscle fibers are not working at their optimal length of the force-length relation, thereby contributing to diaphragm weakness.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Symptoms relating to respiratory or cardiovascular disease
* History of pneumothorax or family history of primary pneumothorax
* Obesity (defined as BMI > 30kg/m²)
* Known pregnancy
* Contraindications for the placement of a nasogastric tube (upper airway/esophageal/gastric/mouth or face pathology (e.g. recent surgery, esophageal varices, diaphragmatic hernia), nasal bleeding within the last 2 weeks or use of anticoagulants)
* Contraindications for MRI (electrical/metallic implants, claustrophobia or history in metalworking)
* Subjects who are employed at the department of intensive care adults, directly involved in the study and/or family from staff of the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in diaphragm's position | 2 hours
  Changes in the position of the diaphragm during different PEEP levels, as measured with both ultrasound and MRI
Changes in diaphragm's shape and length | 2 hours
  Changes of the diaphragm's shape and length during different PEEP levels, as measured with MRI
Changes in diaphragm's efficiency | 2 hours
  Changes in the neuro-mechanical efficiency of the diaphragm (ratio between pressure and electrical muscle activity) during different PEEP levels, as measured with a nasogastric catheter
Change in twitch transdiaphragmatic pressures | 2 hours
  Twitch transdiaphragmatic pressures during different PEEP levels, as measured with magnetic stimulation of the phrenic nerves.

SECONDARY OUTCOMES:
Difference between MRI and ultrasound | 2 hours
  The difference between diaphragm parameters obtained by ultrasound and parameters obtained by MRI

OTHER OUTCOMES:
Expiratory abdominal muscle activity | 2 hours
  Expiratory abdominal muscle activity during different levels of PEEP measured with surface EMG electrodes
Flow | 2 hours
  Flow during different levels of PEEP measured by the non-invasive ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Leo Heunks, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided